CLINICAL TRIAL: NCT01577095
Title: A Randomized Controlled Trial Evaluating the Effects of Electroacupuncture and Rosiglitazone Combined Therapy on Patients With Type 2 Diabetes Mellitus
Brief Title: Evaluating the Effects of Electroacupuncture and Rosiglitazone Combined Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMR94-IRB-139
Record Dates: First submitted 2012-03-27; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus With Features of Insulin Resistance
Keywords: electroacupuncture; rosiglitazone; plasma glucose; insulin resistance; free fatty acid
MeSH Terms: conditions — Insulin Resistance | interventions — Rosiglitazone; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EA + Rosiglitazone (Experimental)
  Interventions: Other: EA + Rosiglitazone
- Rosiglitazone (Placebo Comparator)
  Interventions: Drug: TZD

INTERVENTIONS:
Other: EA + Rosiglitazone — electroacupuncture and Rosiglitazone combined therapy on patient of type II DM
  Other Names: Electroacupuncture and Rosiglitazone combined therapy
  Arms: EA + Rosiglitazone
Drug: TZD — Rosiglitazone 8 mg single dose
  Other Names: The effect of hypoglycemia and improving insulin sensitivity
  Arms: Rosiglitazone

SUMMARY:
Aims: To evaluate the efficacy of rosiglitazone (TZD) and electroacupuncture (EA) combined therapy on patients with type 2 diabetes mellitus (T2DM). A randomized single-blind placebo controlled clinical trial was used.

Methods: A total of 31 newly diagnostic type 2 diabetic patients, who fulfilled the eligibility criteria were recruited and received various allocated interventions. They were randomly assigned into two groups, the control group (TZD, N=15) and the experimental group (TZD + EA, N=16). Changes in their plasma free fatty acid (FFA), glucose and insulin levels together with their homeostasis model assessment (HOMA) indices were statistically assessed between before and after treatment. Hypoglycemic activity (%) was also compared between these two groups.

Expecting Results: This study will compare the hypoglycemic activity and the ability of improving insulin resistance between the TZD and TZD+EA group. Also, the lowering effect of the plasma FFA concentration will be investigated.

DETAILED DESCRIPTION:
This study is compared the effect between combined therapy (EA+TZD) and drug (TZD) on the patient of type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* all included native Taiwanese patients, age from 20 to 65 years who diagnosed with type 2 diabetes mellitus within 5 years and keep the same anti-hyperglycemic agents for control diabetes before and during the period in this study
* compatible with the diagnostic criteria of diabetes mellitus according to American Diabetes Association

Exclusion Criteria:

* individuals with nephrotic syndrome (urine protein over 3.5 g/day) and edema or renal failure (serum creatinine over 115 μmol/L)
* individuals who were diagnosed of heart failure (NYHA Fc III~IV) or pacemaker implantation
* individuals with abnormal liver function (GOT and GPT level above 2 folds of normal range) or diagnosis of liver cirrhosis
* individuals with higher HbA1C level (HbA1C above 9%)
* pregnant women
* individuals who were receiving the classes of drugs thiazolidinediones already
* individuals who were receiving insulin therapy already
* individuals who were receiving other therapy during the period of study
* individuals suffering a homeostasis disorder or other systemic disease
* individuals who did not comply with the treatment during the study period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
plasma glucose | Time point(s) at which outcome measure is assessed in one year
  The primary endpoint with respect to plasma glucose level after treatment in each group of patients and compare the hypoglycemic activity between these two independent groups.

SECONDARY OUTCOMES:
plasma free fatty acid (FFA) | Time point(s) at which outcome measure is assessed in one year.
  This secondary endpoint will compare the percent change of plasma FFA level between these two independent groups.
plasma insulin | Time point(s) at which outcome measure is assessed in one yease
  This secondary endpoint will compare the plasma insulin level after treatment of each group and the change between these two independent groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Liang Chang, PhD, Principal Investigator — China Medical University, China
Locations (1):
- Department of Integrative Chinese-Western Clinic, China Medical University Hospital, Taichung, Taiwan, Taiwan

REFERENCES:
- [Background] Pai HC, Tzeng CY, Lee YC, Chang CH, Lin JG, Cheng JT, Chang SL. Increase in plasma glucose lowering action of rosiglitazone by electroacupuncture at bilateral Zusanli acupoints (ST.36) in rats. J Acupunct Meridian Stud. 2009 Jun;2(2):147-51. doi: 10.1016/S2005-2901(09)60047-9. PMID 20633486
- [Derived] Lin RT, Pai HC, Lee YC, Tzeng CY, Chang CH, Hung PH, Chen YI, Hsu TH, Tsai CC, Lin JG, Chang SL. Electroacupuncture and rosiglitazone combined therapy as a means of treating insulin resistance and type 2 diabetes mellitus: a randomized controlled trial. Evid Based Complement Alternat Med. 2013;2013:969824. doi: 10.1155/2013/969824. Epub 2013 Jul 29. PMID 23983807